CLINICAL TRIAL: NCT01101646
Title: A Phase 1, Open-Label, Randomized, Crossover Study to Assess the Relative Bioavailability of Rabeprazole Phase 3 Pediatric Bead Formulation Versus the Phase 1 Pediatric Bead Formulation and Effect of Food on the Pharmacokinetics of Rabeprazole Phase 3 Pediatric Bead Formulation in Healthy Subjects
Brief Title: A Pharmacokinetic and Relative Bioavailability Study With Rabeprazole Sodium in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CR014827; RABGRD1006
Record Dates: First submitted 2010-03-11; First posted 2010-04-12 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Gastroesophageal Reflux
Keywords: Rabeprazole sodium; Pharmacokinetics; Biological Availability; Safety; Adult
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole

ARMS (3):
- 001 (Experimental): rabeprazole sodium four 2.5 mg capsules of the phase 3 pediatric bead formulation suspended in a strawberry flavored vehicle (taken in fasted or fed state)
  Interventions: Drug: rabeprazole sodium
- 002 (Experimental): rabeprazole sodium two 5-mg sachets of the phase 1 pediatric bead formulation suspended in a strawberry flavored vehicle (taken in fasted state)
  Interventions: Drug: rabeprazole sodium
- 003 (Experimental): rabeprazole sodium four 2.5 mg capsules of the phase 3 formulation sprinkled on 1 ounce of plain yogurt
  Interventions: Drug: rabeprazole sodium

INTERVENTIONS:
Drug: rabeprazole sodium — four 2.5 mg capsules of the phase 3 pediatric bead formulation suspended in a strawberry flavored vehicle (taken in fasted or fed state)
  Arms: 001
Drug: rabeprazole sodium — two 5-mg sachets of the phase 1 pediatric bead formulation suspended in a strawberry flavored vehicle (taken in fasted state)
  Arms: 002
Drug: rabeprazole sodium — four 2.5 mg capsules of the phase 3 formulation sprinkled on 1 ounce of plain yogurt
  Arms: 003

SUMMARY:
The purpose of the study is to evaluate and compare the pharmacokinetics (blood levels) of 2 different formulations, assess the effect of food on the pharmacokinetics and assess safety of rabeprazole sodium in healthy volunteers. Rabeprazole sodium is a drug used to treat patients with Gastro Esophageal Reflux Disease (GERD). GERD is a condition in which the esophagus (tube from throat to stomach) becomes irritated or inflamed because of acid backing up from the stomach.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), open-label (the patient knows the treatment/drug they are taking), single-dose, 3-way crossover study to evaluate and compare the pharmacokinetics (blood levels) and safety of 2 formulations of orally (by mouth) administered rabeprazole sodium in healthy volunteers. Rabeprazole sodium is a drug used to treat patients with Gastro Esophageal Reflux Disease (GERD), a condition in which the esophagus (tube from throat to stomach) becomes irritated or inflamed because of acid backing up from the stomach. The primary outcome measure of the study is to evaluate the relative bioavailability (the rate and extent at which the drug is absorbed and reaches blood circulation ) of rabeprazole sodium (Phase 3 versus Phase 1 formulation) and the effect of food (Phase 3 formulation) by estimation of standard plasma PK parameters (Cmax, the maximum concentration of the drug in the blood observed after its administration; tmax, the time it takes for the drug to reach its maximum concentration in the blood after its administration; and AUC [the area under the curve]) of rabeprazole and its major metabolite.Blood samples to assess the PK of study drugs will be obtained before and up to 16 hours after dosing on Day 1 during 3 treatment periods. Thirty-six (36) healthy volunteers will be enrolled and will participate in the study for a total of approximately 36 days (from beginning of screening until the end-of-study procedures). During the study, the healthy volunteer will make a total of approximately 4 visits to the study center. The 4 visits will include a screening visit and three 2-day inpatient stays to receive study drug. During the screening visit, the details regarding the study will be explained and if the volunteer wishes to participate in the study, a signed informed consent form will be obtained. After informed consent is obtained, study specific entry criteria will be reviewed with the volunteer, information regarding the volunteer's medical history and demographics (age, race, etc) will be collected, and the following procedures will be performed: physical examination, measurement of vital signs (pulse rate and blood pressure), 12-lead electrocardiogram (ECG), serum pregnancy test (for women of childbearing potential), serology, drug screen and alcohol test, and laboratory testing (hematology, serum chemistry, and urinalysis). During each treatment period, volunteers who fulfill study enty criteria will be randomized to receive 1 of 3 treatments as follows: (1) a strawberry flavored suspension of the phase 1 formulation of study drug in a fasted state (2) a strawberry flavored suspension of the phase 3 formulation of study drug in a fasted state , and (3) a strawberry flavored suspension of the phase 3 formulation of study drug in a fed state (with food) OR phase 3 formulation of study drug sprinkled on 1 ounce of plain yogurt. During each 2-day treatment period, volunteers will be admitted to the study center after an overnight fasting (withholding consumption of food) period of at least 8 hours before blood is drawn for laboratory safety testing on Day 1, receive study drug on Day 1, and remain overnight at the study center unit for completion of all Day 2 study procedures. After all Day 2 study procedures are completed, the volunteer will be discharged from the study center unit for a 7- to 14-day period and then return to the study center for the 2nd treatment period. The same procedures will be followed for treatment periods 2 and 3. During the study, safety will be monitored by the measurement of vital signs before and after dosing during each treatment period, ECG findings at screening and at the end-of-study (Day 2 of treatment period 3 or at the time of early withdrawal from the study), and the evaluation of adverse events reported from the time of screening through to the end of the study. In each of 3 treatment periods, healthy volunteers will receive the equivalent of a 10 mg dose of rabeprazole sodium (ie, four 2.5 mg capsules of the phase 3 pediatric bead formulation or two 5-mg sachets of the phase 1 pediatric bead formulation) mixed with a strawberry-flavored vehicle and administered orally as a suspension or they will receive four 2.5 mg capsules of the phase 3 formulation sprinkled on plain yogurt to be ingested (eaten).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer with no clinically relevant abnormalities as determined by medical history, physical examination, blood chemistry, hematology, urinalysis, vital signs, and electrocardiogram (ECG)
* Agrees to abstain from alcohol intake 48 hours before each study drug administration and during the inpatient portions of the study
* Agrees not to consume food containing poppy seeds during the study or food/beverages containing grapefruit juice, seville oranges, or quinine (eg, tonic water) from 72 hours prior to Study Day -1 until after the last PK sample is collected
* Agrees to limit intake of caffeine/methylxanthine (eg, coffee, tea, chocolate, or caffeine-containing soft drinks) to less than 300 mg/day (eg, approximately 3 cups of coffee or 6 cola drinks) for the duration of the study
* Female volunteers of childbearing potential agree to use appropriate birth control method during the study

Exclusion Criteria:

* Currently have, or have a history of disease or dysfunction of the pulmonary, cardiovascular, endocrine, hematologic, neurological, immune, gastrointestinal, genitourinary, or other body system that is clinically significant in the opinion of the Investigator
* Have evidence of any chronic medical conditions requiring prescription medications
* History of hypersensitivity or allergies to any drug compound, including rabeprazole sodium, substituted benzimidazoles, or any excipient used in pediatric bead formulation, unless approved by the Investigator
* Have had major or traumatic surgery within 12 weeks prior to screening or pre-planned surgery or procedures that would interfere with the conduct of the study
* Have an acute illness within 7 days prior to study drug administration or have had a major illness or hospitalization within 1 month prior to study drug administration
* Have a recent history (within previous 1 year) of alcohol or drug abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the relative bioavailability of rabeprazole sodium (Phase 3 versus Phase 1 formulation) and the effect of food (Phase 3 formulation) by estimation of standard plasma PK parameters (Cmax. AUC, tmax) of rabeprazole and its major metabolite. | Before and up to 16 hours after study drug administration on Day 1 during treatment periods 1, 2, and 3

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of 2 formulations of rabeprazole sodium by assessment of vital signs, clinical laboratory tests, physical examinations, ECG findings, and adverse events. | Approximately 36 days (includes time of screening through to the end of the study or early withdrawal)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Overland Park, Kansas, United States

REFERENCES:
- [Derived] Thyssen A, Solanki B, Gonzalez M, Leitz G, Treem W, Mannaert E. Pharmacokinetics of rabeprazole granules versus tablets, and the effect of food on the pharmacokinetics of rabeprazole granules in healthy adults-cross-study comparison. Clin Pharmacol Drug Dev. 2014 Sep;3(5):406-16. doi: 10.1002/cpdd.118. Epub 2014 May 23. PMID 27129014